CLINICAL TRIAL: NCT05105087
Title: Detection of Sentinel Lymph Nodes in Female Lower Genital Tract Cancer Patients With Contrast-Enhanced Ultrasound Imaging
Brief Title: Gynecological Sentinel Lymph Nodes CEUS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21F.624; R21CA249870 (NIH); JT 16886 (Other: JeffTrial Number)
Record Dates: First submitted 2021-08-13; First posted 2021-11-03 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Cervical Carcinoma; Malignant Female Reproductive System Neoplasm; Vaginal Carcinoma; Vulvar Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms | interventions — Sonazoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (perflubutane microbubble, ultrasound) (Experimental): Patients receive perflubutane microbubble injections subdermally and then undergo ultrasound over 30 minutes before standard of care cancer treatment.
  Interventions: Drug: Perflubutane Microbubble; Procedure: Contrast-Enhanced Ultrasound

INTERVENTIONS:
Drug: Perflubutane Microbubble — Given subdermally
  Other Names: Sonazoid; gas-filled microbubbles
Procedure: Contrast-Enhanced Ultrasound — Undergo ultrasound
  Other Names: CEUS

SUMMARY:
This clinical trial compares the use of ultrasound for the detection of sentinel lymph nodes (SLNs) to the standard of care (which varies depending on cancer treatment). The ultrasound contrast agent is called Sonazoid and it consists of tiny gas-filled bubbles about the side of red blood cells. Diagnostic procedures, such as ultrasound with Sonazoid, may help identify more SLNs than standard of care in patients with cervical, vaginal, or vulvar cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the concordance between lymphosonography and the standard of care in the identification sentinel lymph nodes (SLNs) in patients with cervical, vaginal or vulvar cancer.

II. To determine if lymphosonography can identify more SLNs with metastatic deposits in patients with cervical, vaginal or vulvar cancer when compared to the standard of care.

OUTLINE:

Patients receive perflubutane microbubble (Sonazoid) injections subdermally and then undergo ultrasound over 30 minutes before standard of care cancer treatment.

After completion of study intervention, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Be female
* Be diagnosed with cervical, vaginal or vulvar cancer
* Be at least 18 years of age
* If of child-bearing potential, must have a negative pregnancy test
* Be able to comply with study procedures
* Have read and signed the Institutional Review Board (IRB)-approved informed consent form for participating in the study

Exclusion Criteria:

* Females who are pregnant or nursing
* Patients who have received an investigational drug in the 30 days before study drug administration, or will receive one within 72 hours afterwards
* Patients who are medically unstable, patients who are seriously or terminally ill, and patients whose clinical course is unpredictable. For example:

  * Patients on life support or in a critical care unit
  * Patients with clinically unstable cardiac arrhythmias, such as recurrent ventricular tachycardia
  * Patients with recent cerebral hemorrhage
  * Patients who have undergone surgery within 24 hours prior to the study sonographic examination
* Patients with congenital heart defects
* Patient with a known allergy to Sonazoid (including an anaphylactic allergy to eggs or egg products)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2025-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Bin Liu, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-site, open-label, non-randomized pilot study conducted at Thomas Jefferson University (TJU), Sidney Kimmel Cancer Center, Philadelphia, PA. Subject recruitment was expected to last 24 months, beginning in April 2022 and ending in November 2023. Recruitment was conducted from the patient population of the Department of Gynecology Oncology at TJU. Eligible participants were identified by surgical co-investigators from their existing patient population.
Pre-assignment Details: Screening assessments were performed within 4 weeks prior to the administration of Sonazoid. A full demographic profile, known drug allergies or intolerances, and a review of the subject's medical/surgical history were recorded.
  9 participants received CEUS. 5 completed both CEUS and surgery with pathology and were analyzed. 2 were ineligible for surgery (advanced disease), and 2 withdrew consent prior to surgery; thus no outcome data were available for these 4 participants.
Period: Overall Study
Arm/Group | Diagnostic (Perflubutane Microbubble, Ultrasound)
Started | 9
Completed | 5
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Ineligible for surgery due to advanced disease | 2

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (Perflubutane Microbubble, Ultrasound)
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants] — Population: Only patients who completed both CEUS and surgery with SLN excision and pathology evaluation (N=5) were included for analysis.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 4
    >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 55 [36 to 75]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only patients who completed both CEUS and surgery with SLN excision and pathology evaluation (N=5) were included for analysis.
  Participants
    Female | 5
    Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only patients who completed both CEUS and surgery with SLN excision and pathology evaluation (N=5) were included for analysis.
  Participants
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 3
    White | 1
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Sentinel Lymph Nodes (SLNs) Identified by Lymphosonography as Well as Blue Dye or Positron Emission Tomography (PET)-Computed Tomography (CT)
Description: The number of SLN detected by contrast enhanced ultrasound will be compared to the number of SLN detected by the standard of care (i.e., by blue dye or by PET-CT).
Time Frame: up to 30 minutes during CEUS procedure
Population: Only participants who completed CEUS and surgery (N=5) were analyzed.
Measure: Number; unit: sentinel lymph nodes (SLNs)
Units Other Than Participants: sentinel lymph nodes (SLNs)
Arm/Group | Diagnostic (Perflubutane Microbubble, Ultrasound)
Number analyzed (Participants) | 5
Number analyzed (sentinel lymph nodes (SLNs)) | 17
sentinel lymph nodes (SLNs) | 17

2. Secondary Outcome: Location of Sentinel Lymph Nodes (SLNs) Identified by Contrast-enhanced Ultrasound (CEUS)
Time Frame: up to 30 minutes during CEUS procedure
Population: Only participants who completed CEUS and surgery (N=5) were analyzed.
Measure: Number; unit: sentinel lymph nodes (SLNs)
Units Other Than Participants: sentinel lymph nodes (SLNs)
Arm/Group | Diagnostic (Perflubutane Microbubble, Ultrasound)
Number analyzed (Participants) | 5
Number analyzed (sentinel lymph nodes (SLNs)) | 17
sentinel lymph nodes (SLNs)
  Left Inguinal Region | 9
  Left Iliac Region | 7
  Right Iliac Region | 1

3. Secondary Outcome: Size of Sentinel Lymph Nodes (SLNs) Identified
Description: The locations, depth beneath the skin surface and size (measured in three orthogonal dimensions) of each SLN will be recorded.
Time Frame: up to 30 minutes during CEUS procedure
Population: Only participants who completed CEUS and surgery (N=5) were analyzed.
Measure: Mean (Full Range); unit: centimeters (cm)
Units Other Than Participants: sentinel lymph nodes (SLNs)
Arm/Group | Diagnostic (Perflubutane Microbubble, Ultrasound)
Number analyzed (Participants) | 5
Number analyzed (sentinel lymph nodes (SLNs)) | 17
centimeters (cm) | 1.6 [0.7 to 2.4]

4. Secondary Outcome: Depth Beneath the Skin Surface of Each SLN
Description: The locations, depth beneath the skin surface and size (measured in three orthogonal dimensions) of each SLN will be recorded - [this verbiage comes directly from the protocol]
Time Frame: up to 30 minutes during CEUS procedure
Population: Only participants who completed CEUS and surgery (N=5) were analyzed.
Measure: Mean (Full Range); unit: centimeters (cm)
Units Other Than Participants: sentinel lymph nodes (SLNs)
Arm/Group | Diagnostic (Perflubutane Microbubble, Ultrasound)
Number analyzed (Participants) | 5
Number analyzed (sentinel lymph nodes (SLNs)) | 17
centimeters (cm) | 2.71 [0.5 to 6.0]

5. Secondary Outcome: Presence of Metastatic Deposits in the Sentinel Lymph Node (SLNs)
Description: The presence or absence of metastatic deposits in SLNs will be obtained by pathology (when available).
Time Frame: Within 7 days post-surgery
Population: Only participants who completed CEUS and surgery (N=5) were analyzed.
Measure: Number; unit: Metastatic sentinel lymph nodes (SLNs)
Units Other Than Participants: sentinel lymph nodes (SLNs)
Arm/Group | Diagnostic (Perflubutane Microbubble, Ultrasound)
Number analyzed (Participants) | 5
Number analyzed (sentinel lymph nodes (SLNs)) | 11
Metastatic sentinel lymph nodes (SLNs) | 3

ADVERSE EVENTS:
Time Frame: The PI will follow AEs with start dates occurring any time after informed consent is obtained until 7 (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation. Events will be followed for outcome information until resolution or stabilization.
Arm/Group | Diagnostic (Perflubutane Microbubble, Ultrasound)
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT05105087/Prot_SAP_000.pdf